CLINICAL TRIAL: NCT00539630
Title: TAX + Cisplatin + 5 F/U vs Cisplatin + 5 F/U in SCCHN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976F_3501
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Last update posted 2007-10-04 (Estimated); Status verified 2007-10

CONDITIONS: Carcinoma, Squamous Cell
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Docetaxel

INTERVENTIONS:
Drug: Docetaxel

SUMMARY:
To describe the clinical response rate in two groups (Docetaxel plus cisplatin plus 5-FU, versus Cisplatin plus 5-FU) after 3 cycle of neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven squamous cell carcinoma of the head and neck with locally advanced inoperable disease.
* Primary tumor sites eligible: oral cavity, oropharynx, hypopharynx , larynx or nasopharynx.
* Patients are required to have at least one (bi-or uni-dimensionally) measurable lesion.
* WHO performance status 0 or 1.
* Adequate bone marrow, hepatic and renal functions.

Exclusion Criteria:

* Pregnant and lactating women
* Previous chemotherapy
* Previous radiotherapy for H&N
* Previous surgery for H&N

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2002-11

PRIMARY OUTCOMES:
Clinical response will be evaluated by modified WHO criteria. Clinical and radiological assessment of all lesions will be performed | After 2 cycle, 3 cycle and after concurrent chemo/radiotherapy.

SECONDARY OUTCOMES:
Pathologic response if clinical response of primary tumor is CR at the end of chemotherapy and end of concurrent chemo/ radiotherapy, biopsy of primary tumor site will be performed to evaluate pathologic response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Hyang Rim Kim, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Seoul, South Korea